CLINICAL TRIAL: NCT03145168
Title: High Versus Low Target Mean Arterial Pressure in Septic Shock in Critically Ill Cirrhotics -A Randomized Controlled Trial
Brief Title: High Versus Low Target Mean Arterial Pressure in Septic Shock in Critically Ill Cirrhotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-08
Record Dates: First submitted 2017-04-10; First posted 2017-05-09 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Target Mean Arterial Pressure (Experimental)
  Interventions: Other: High Target Mean Arterial Pressure
- Low target Mean Arterial Pressure (Active Comparator)
  Interventions: Other: Low Target Mean Arterial Pressure

INTERVENTIONS:
Other: High Target Mean Arterial Pressure — High target group (80-85 mm of Hg).
  Arms: High Target Mean Arterial Pressure
Other: Low Target Mean Arterial Pressure — Low target MAP group (60-65mm Hg).
  Arms: Low target Mean Arterial Pressure

SUMMARY:
Study Design:

* A randomized controlled study.
* The study will be conducted on patients admitted to Department of Hepatology from April 2017 to October 2017 at ILBS, New Delhi
* Study group will comprise of patients critically ill cirrhotics with septic shock

All included patients would be randomised to low target MAP group (60-65mm Hg) or high target group (80-85 mm of Hg). Patients older than 18 years of age will be enrolled if they have septic shock that is refractory to fluid resuscitation and if they required vasopressors (norepinephrine or epinephrine or terlipressin) at a minimum infusion rate of 0.1 μg per kilogram per minute. Standard criteria will be considered to define refractoriness to fluids. The target MAP would be maintained for a max. of 5 days or until recovery or shock and or AKI. In the high-target group, a reduction in vasopressor doses to maintain a mean arterial pressure of 65 to 70 mm Hg will be done in case of any of the prespecified serious adverse events that could potentially be related to an increased rate of vasopressor infusion occurred. These events could be: clinically relevant bleeding (i.e., transfusion requirements of at least 2 units of packed red cells), myocardial infarction (defined as typical electrocardiographic changes, with a concomitant increase in troponin, and segmental echocardiographic hypokinesia or akinesia, with the infarction confirmed, when possible, by means of coronary angiography), major ventricular arrhythmia, poorly tolerated supraventricular arrhythmia, mesenteric ischemia, and distal-limb ischemia.

• Septic shock would be defined as clinical construct of sepsis with persisting hypotension requiring vasopressors to maintain MAP>=65 mm of Hg and having a serum lactate >2 mmol/L despite adequate volume resuscitation

ELIGIBILITY:
Inclusion Criteria:

* Critically ill cirrhotics with septic shock

Exclusion Criteria:

* Patients with age less than 18 years
* Severe known cardiopulmonary disease (structural or valvular heart disease, coronary artery disease, COPD)
* Pregnancy
* Chronic kidney disease on hemodialysis
* Extremely moribund patients with an expected life expectancy of less than 24 hours
* Failure to give informed consent from family members.
* Hemodynamic instability requiring very high dose of vasopressors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
Survival in both groups | 28 days

SECONDARY OUTCOMES:
Duration of mechanical ventilation | 3 months
Incidence of intradialytic hypotension in patients undergoing Renal Replacement Therapy | 3 months
Duration of Intensive Care Unit /Hospital stay | 3 months
Reversal of shock in both groups | Day 5
Acute Kidney Injury in both groups. | Day 5

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maiwall R, Rao Pasupuleti SS, Hidam AK, Kumar A, Tevethia HV, Vijayaraghavan R, Majumdar A, Prasher A, Thomas S, Mathur RP, Kumar G, Sarin SK. A randomised-controlled trial (TARGET-C) of high vs. low target mean arterial pressure in patients with cirrhosis and septic shock. J Hepatol. 2023 Aug;79(2):349-361. doi: 10.1016/j.jhep.2023.04.006. Epub 2023 Apr 23. PMID 37088310